CLINICAL TRIAL: NCT04886947
Title: "Use of Autologous Umbilical Cord Stem Cell Transplantation in the Reconstruction of Alveolar Cleft "
Brief Title: Alveolar Cleft Reconstruction Powered by
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAKRIF/DVCFA/025/20
Record Dates: First submitted 2021-05-11; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Alveolar Cleft
Keywords: alveolar cleft stem cell gingivoperiosteoplasty
MeSH Terms: interventions — Stem Cell Transplantation

STUDY DESIGN:
Intervention Model Description: case control study with control being those receiving convectional treatment and cases those will have added intervention of autologues stem cell
Masking Description: The radiologist interpreting bone formation of the alveolar will be blinded on which group the participants belongs. whether no or intervention done
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stem cell intervention (Experimental): Arm A patients who will have surgery with stem cell added.
  Arm B only surgery with no stem cell added.
  Interventions: Procedure: stem cell transplantation

INTERVENTIONS:
Procedure: stem cell transplantation — After surgical repair of alveolar cleft using gingivoperiosteoplasty, processed and stored autologous stem cells will be added at the repair site. After which the patient will be followed up for bone regeneration and this will be compared to control where no stem cell is added.

SUMMARY:
More than four million children are born with birth defects worldwide every year and a million presenting with cleft lip and palate. Cleft lip and palate is a congenital defect of the lip alveolar and palate it's now recognized as a significant cause of infant mortality and childhood morbidity and included among global burden of disease initiative. In Uganda the estimated number of babies born with cleft lip and palate is 1100 per year Children with 75% of them having alveolar cleft which is a defect in the upper jaw (Maxilla arch).

The secondary bone graft and gingivoperiosteoplasty have become the two popular approaches to bone generation in alveolar defect. These two methods have varying success rates; primary gingivoperiosteoplasty 50 to 60% and secondary bone graft is 87% but Gingivoperiosteoplasty is the preferred option to many African surgeons to obviate the need for bone grafting which is technically demanding, prolonging therapy with many procedures therefore poor compliance, also increasing treatment failure rate and has significant associated donor morbidity. This project is set out to address the challenge of bone regeneration in alveolar cleft and improve on the surgical outcome by the use of stem cell therapy.

The objective of this study is to compare the outcome of umbilical cord blood stem cell transplant plus gingivoperiosteoplasty to conventional gingivoperiosteoplasty on timing and density of bone regeneration.

1.3. Hypothesis In this study we hypothesize that primary repair with gingivoperiosteoplasty the success rate can be improved or enhanced with the use of stem cell therapy in our setting.

Alternative hypothesis: Autologous umbilical stem cells transplantation following gingivoperiosteoplasty results in better bone regeneration when compared to gingivoperiosteoplasty.

Null hypothesis: Autologous umbilical stem cells transplantation following gingivoperiosteoplasty has no benefit on promoting bone regeneration when compared to gingivoperiosteoplasty alone.

The study will be a case control pilot study conducted in Kiruddu National Referral hospital Kampala Uganda. 20 participants who will be neonates of either sex with unilateral cleft lip and palate will be recruited in the study. They will be split into two groups: group A will have the umbilicus cord and placenta blood collected at birth and group B will not have umbilical cord or placenta blood collected and will be designated as the Control group.

DETAILED DESCRIPTION:
A lot has progressed in the care of Cleft lip and palate with development of multidisciplinary team approach. Despite these achievements there are still a lot of challenges in the treatment of alveolar cleft. Alveolar cleft being the less conspicuous component of the cleft abnormality attracted less interest in its correction; its treatment history dates in the not-so-distant past were as cleft lip history repair dates as far as 390 Before Christ and palate repair in 1764. The first attempt to treat alveolar cleft with bone graft was in 1901 then again in 1908 but it was not until 1914 that Dracher was the first to perform a successful bone graft of the alveolar defect using tibial bone that gave birth to the primary alveolar bone graft. This approach was later found to be destructive to the developing face and was abandoned. Then in 1972 Secondary bone grafting of maxilla and residual alveolar clefts at the stage of transitional dentition this become popular in some centers.

In 1967 Swedish Plastic Surgeon Tord Skoog introduced yet a new concept called boneless alveolar graft or primary periosteoplasty (PPP) which he performed during the time of lip repair at 3 months in this repair periosteal flaps were raised clearing soft tissue between the alveolar defect and the flaps were closed to form a tunnel at the time of lip repair. This was because it was believed that with time bone would form in the tunnel and so bone graft will not be needed. Follow up in many studies indicated bone developed in the tunnel in about 60 to 72% of the cases. His follow up study up to the age of 18years indicated that despite a delay in facial growth at early age by 18 years all are at the same level.

This study is set out to address the challenge of bone regeneration in alveolar cleft and improve on the surgical outcome by the use of stem cell therapy in African population. All the documented studies are conducted only in non-African populations which have slightly different phenotype and use to pre-surgical orthodontic treatment.

Stem-cells are un-differentiated progenitor cells capable of self-renewal and differentiation into any specialized cells. Umbilical cord stem cells in gingivoperiosteoplasty has shown good bone regeneration in alveolar cleft and minimizing the donor mobility. But there is a need for us to establish its possibility and effectiveness in out setting. This will be the first stem cell trial in cleft treatment protocol in our region . With the establishment of a stem cell center at Makerere and recently funded to improve its capacity, we believe we can contribute to the improvement of cleft care in Uganda.

Problem statement The current accepted gold standard protocol for alveolar defect is controversial on timing, outcome, and associated morbidity. Therefore, the second common protocol of Gingivoperiosteoplasty (GPP) carried out during primary lip repair at 3 to 6 months would provide a better alternative by providing early repair with a smaller number of surgeries and also obviate the need for secondary bone graft with further use of stem cell transplant. The use of umbilical stem cell transplantation in gingivoperiosteoplasty procedure has only been done in 10 cases and the results indicate good bone regeneration in the alveolar bone defect. Despite the demonstration of success in the previous stem cell therapy there is need to do a clinical trial in African population to prove the role and use of stem cells in alveolar bone regeneration in our setting.

Significance The findings of this study will demonstrate the therapeutic role of stem-cell therapy as an effective alternative bone generator to bone graft in correction of alveolar defect in cleft lip and palate. This will present a paradigm shift in the treatment of patients with cleft lip and palate by eliminating the need for secondary bone graft. Such a study will also promote the establishment by Makerere University and the government of super-specialized treatment such as stem-cell therapy. closing the gap between academia stem cells in the laboratory and clinical practice. This study currently being the only clinical trial in the use of umbilical blood stem in alveolar reconstruction in the region will pave way for further utilization of stem cells as well as developing standard operating procedures.

1.6. Justification The theory of GPP is consistent with the goal of minimizing the number of secondary surgeries by optimizing results of primary surgery. And the most important outcome obtained is the elimination of secondary bone graft. It's important to have limited dissection to prevent risk of iatrogenic restriction of facial growth so introduction of an additional source of bone generation will further improve on the outcome of GPP with no need for extensive dissection. This study will also improve on the knowledge attitude and practice of the use of umbilical cord blood stem cells for clinical purpose and more so in surgery to generate bone. The umbilical cord stem cell is chosen as the source of stem cells because it has a high number and high rate of regeneration Being the first study in our setting on primary alveolar repair we propose the finding will define the role of stem cell therapy in cleft lip and palate surgery and demonstrate the usefulness of stem cells in the future of correcting alveolar defect with no need of bone graft.

2.2. STUDY PROCEDURE We shall establish a surveillance team in Mulago Women's hospital, Kawempe and Mukono Hospital Plus Kisenyi health center. The Ante Natal Care radiology team in these centers will be trained on the key parameters of interest and once they identify any fetus with a cleft lip and palate on ultrasound, they will obtain the mothers demographics including the phone contact. Once this information is provided to the PI, the mothers will be contacted and evaluated for eligibility. In case they meet the preliminary eligibility criteria, informed consent will be obtained and the mothers will be followed up to the time of delivery.

If the child born has unilateral cleft lip and cleft palate with clinical evidence of alveolar cleft will be recruited into the study and then placenta and cord blood will be collected for harvest of stem cells will be known the cases: A arm Arm B: Children with cleft lip and palate having similar clinical presentation of cleft lip and palate where it was not possible to collect umbilical cord and placental blood will be the Control group.

The surgical procedure will be done by a single plastic surgeon and the same surgical technique for all participants.

Stem cell group mothers will have screening for HIV, Hepatitis done before processing of the stem cell if found reactive the process will not proceed.

Interventional arm A:

Collection of Umbilical cord blood:

• Umbilical cord blood will be collected by midwives using Marcopharma Cord blood collection kit (https://www.macopharma.com/products/collection-bags/) (figure #). Once the baby is safely delivered, the midwife will clamp the umbilicus end near the baby and add another clamp two centimeter above and a transection made between both clamps after appropriately disinfecting. Using the collection bag set, a needle will be inserted into the vein in the cord and blood allowed to flow by gravity into the bag. When the flow stops, the blood bag will be clamped to prevent leakage and the bag gently inverted for 8 to 10 times to allow normal mixing with the anticoagulant. The bag will then be labeled with the unique patient ID and mother's details, collection tubing arm clipped and the bag sealed. The bag will then be placed in a biohazard ziplock bag labeled with the mother's details and then placed in a cool box at room temperature. And transported to the laboratory.

Processing of the stem cells:

• Once the cord blood collection bags and tissue reach the laboratory, any tubing attached to the bag will be stripped and mix very thoroughly ensuring that the tubings are sealed. The stem cells will be processed and prepared for cryopreservation.

Cryopreservation of stem cells:

* The density of cells required for Cryopreservation will be determined based on the cell count results as this will help determine the volume of Cryopreservation Medium needed.
* Cells will be suspended in the cryopreservation medium and centrifuged at 200 x g for 10 min. And the media aspirated, leaving behind the cell pellet.
* The cell pellet will be resuspended in the appropriate volume of the cryopreservation medium.
* Suspended cells will be transferred into sterile cryovials.
* Once the cell suspension has been transferred to a sterile cryovial, the cryovial will be transferred to a -80°C freezer and stored vertically for a 24-hr. time period.
* At the end of 24 hrs., the tubes will be transferred into a liquid nitrogen storage unit for long-term cryostorage.

Thawing and preparation for infiltration:

* 2 wells of Matrigel will be prepared the day before thawing the cells.
* Cells will be thawed quickly by swirling the vial in a 37oC water bath until only a small chip of frozen material remains.
* The vial will be swabbed with alcohol and place in the tissue culture hood and the contents transferred to a 15ml tube
* 5ml of pre-warmed culture medium will be added and mixed gently.
* If there are many visible colonies, they will be allowed to sediment at room temperature for 5 min. If colonies are not visible, spin at 200g for 5 min.
* The supernatant will be aspirated and resuspended in 2ml of culture medium.
* 1 well of Matrigel will be aspirated and thawed cells added to it.
* Colonies will evenly be distributed by gentle agitation and incubate overnight in a tissue culture incubator (37oC/5% CO2).
* The next day, the second well of Matrigel will be aspirated and the supernatant transferred from the first well onto it and 2ml of culture medium will be added.
* The colonies will be evenly distributed by gentle agitation and incubated overnight in a tissue culture incubator (37oC/5% CO2).

2.2.2.1.5. Interventional Arm A; Surgical procedure:

* Cleft and palate repair will be done at 3 to 6 months
* The repair will be done under general anesthesia with vasoconstrictor injection.
* Osseus tunnel will be created by removing soft tissue between the 2 alveolar segments.
* The roof of the tunnel will be created using the nasal flaps
* The floor will be created by closure of the oral flaps.
* The anterior lower wall will be created by the labial flaps.
* The anterior superior wall is created with the lip mucosa.
* Thus, the chamber is sealed nasally, orally, and labially by mucoperiosteal flaps

Infiltration of the stem cells:

Stem cells will be injected in and around the tunnel and some of the stem cells will be scuffled in surgicel and placed within the osseus tunnel.

Post infiltration processing and handling:

• Patients will be monitored after surgery for 48 hours to one moth for any complications then at 3 months and 6 months for bone regeneration. Using CT scan.

The control group; We be selected with the same clinical presentation similar age group and having the same surgical procedure except there will be no intervention of stem cell. And also followed from one week to a moth for complications then 3 and 6 months CT scan to monitor alveolar bone growth.

ELIGIBILITY:
Inclusion Criteria:

Neonates with unilateral cleft lip and palate and having clinical evidence of alveolar defect.

Exclusion Criteria:

- Patients with very wide cleft lip and palate Patients whose parents refuse consent Patients with Syndromic cleft

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Alveolar bone density | 6 months
  Alveolar bone density: this will be measured in mm by one radiologist.
Alveolar bone volume | 6 months
  Chelsea scale will be used to score the alveolar bone volume.

OTHER OUTCOMES:
Development of side effects. | one month
  Development of side effects. These will be graded as either Mild: Awareness of a sign or symptom which does not interfere with the participants usual daily activities or is transient and resolves with the use of simple interventions.
  Moderate: Interferes with the participants usual daily activity and required symptomatic treatment including analgesia Severe: Symptoms causing severe discomfort with significant impact of the participant's usual daily activity.
  Serious: Any unexpected medical incident which requires hospitalization or results in long term disability or death.

CONTACTS AND LOCATIONS:
Overall Officials: naknwagi cephas, bachelor, Study Director — Makerere University

IPD SHARING:
Plan to Share IPD: No
there will be no participants data sharing

REFERENCES:
- [Background] Coots BK. Alveolar bone grafting: past, present, and new horizons. Semin Plast Surg. 2012 Nov;26(4):178-83. doi: 10.1055/s-0033-1333887. PMID 24179451
- [Background] Mazzetti MPV, Alonso N, Brock RS, Ayoub A, Massumoto SM, Eca LP. Importance of Stem Cell Transplantation in Cleft Lip and Palate Surgical Treatment Protocol. J Craniofac Surg. 2018 Sep;29(6):1445-1451. doi: 10.1097/SCS.0000000000004766. PMID 30067525
- [Background] Bajestan MN, Rajan A, Edwards SP, Aronovich S, Cevidanes LHS, Polymeri A, Travan S, Kaigler D. Stem cell therapy for reconstruction of alveolar cleft and trauma defects in adults: A randomized controlled, clinical trial. Clin Implant Dent Relat Res. 2017 Oct;19(5):793-801. doi: 10.1111/cid.12506. Epub 2017 Jun 28. PMID 28656723
- [Background] Bhattacharya S, Khanna V, Kohli R. Cleft lip: The historical perspective. Indian J Plast Surg. 2009 Oct;42 Suppl(Suppl):S4-8. doi: 10.4103/0970-0358.57180. PMID 19884680
- [Background] Tanikawa DYS, Pinheiro CCG, Almeida MCA, Oliveira CRGCM, Coudry RA, Rocha DL, Bueno DF. Deciduous Dental Pulp Stem Cells for Maxillary Alveolar Reconstruction in Cleft Lip and Palate Patients. Stem Cells Int. 2020 Mar 12;2020:6234167. doi: 10.1155/2020/6234167. eCollection 2020. PMID 32256610